CLINICAL TRIAL: NCT04083365
Title: A Phase II Study of Capecitabine Plus Concomitant Radiotion Therapy Followed by Durvalumab (MEDI4736) as Preoperative Treatment in Rectal Cancer.
Brief Title: Capecitabine Plus Concomitant Radiation Therapy Followed by Durvalumab as Preoperative Treatment in Rectal Cancer
Acronym: PANDORA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AUSL Romagna Rimini (Other)
Collaborators: AstraZeneca (Industry); Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANDORA
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: RECTAL CANCER
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPECITABINE + concomitant RT + Durvalumab (Experimental): After careful staging, patients will be initiated to a standard concomitant chemoradiation therapy with 825 mg/m2 twice daily capecitabine every day for 5 weeks and 5040 cGy radiotherapy for 5 days per week for 5 weeks. At the end of treatment patients will undergo a lesion biopsy. One week after the end of CT/RT patients will be treated with 1500 mg IV Q4W durvalumab for 3 administrations. From week 9 to 10 after neoadjuvant therapy will be performed re-staging with CT and MRI scan. Surgery will be performed at week 10-12 from the end of CT/RT and the surgical piece will be analyzed
  Interventions: Drug: Capecitabine; Drug: Radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Drug: Capecitabine — chemoradiation therapy with 825 mg/m2 twice daily capecitabine every day for 5 weeks
Drug: Radiotherapy — 5040 cGy radiotherapy for 5 days per week for 5 weeks
Drug: Durvalumab — One week after the end of CT/RT patients will be treated with 1500 mg IV Q4W durvalumab for 3 administrations

SUMMARY:
This is a prospective phase II, open label, single arm, multi-centre study to evaluate activity of an innovative sequence on capecitabine plus concomitant radiation therapy followed by durvalumab in patients with operable rectal cancer. The enrollment period will be of 12 months. Eligible patients will be initiated to a standard concomitant chemoradiation therapy for 5 weeks. One week after the end of CT/RT patients will be treated with durvalumab for 3 administrations. Patient will undergo surgery after 10-12 weeks from the end of CT/RT and the surgical piece will be analyzed. After surgery patients will be followed up for 5 years, according to clinical practice.

ELIGIBILITY:
Inclusion Criteria

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and Data Privacy Directive obtained from the patient/legal representative prior to performing any protocol- related procedures, including screening evaluations.
2. Age > 18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) 0 or 1.
4. Histological diagnosis of adenocarcinoma of rectum.
5. Clinical stage 2-3 rectal adenocarcinoma, cT3/4N0/M0 or Tx N1-2/M0, assessed by thorax abdomen pelvis with contrast Computed tomography (CT) scan, pelvi Magnetic resonance imaging (MRI) scan, pancolonscopy.
6. Able to swallow oral medication.
7. Body weight >30kg.
8. Adequate normal organ and marrow function as defined below:

   1. Haemoglobin ≥9.0 g/dL - Absolute neutrophil count (ANC) > 1500 per mm3
   2. Platelet count >100.000 per mm3
   3. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   4. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
   5. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976).
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre- menopausal patients. Women of childbaring potential or male patients with a female partner of childbearing potential must agree to use at least 1 highly effective method of contraception from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy) as detailed in section 7.1. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   1. Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post- menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up. 11. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Previous treatment for local advanced rectum cancer.
2. Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study. 3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
3. History of hypersensitivity to fluorouracil.
4. Known Dihydropyrimidine dehydrogenase (DPD) deficiency.
5. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease - Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
6. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
7. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
8. Major surgical procedure within 28 days prior to the first dose of treatment.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement - Any chronic skin condition that does not require systemic therapy
    3. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    4. Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of leptomeningeal carcinomatosis.
13. History of active primary immunodeficiency.
14. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
16. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
17. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
18. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
19. Patients unable to follow the Protocol procedures and to sign the informed consent. In the case of patients' incapable of giving informed consent, it must be provided and signed by guardians or legal representative. Patients incapable must also sign the agreement to the extent that they are able to do so.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate after durvalumab treatment | 36 months
  The primary end point will be assessed by means of the proportion of patients having complete pathological response pCR after durvalumab treatment. Corresponding two-sided 95% confidence intervals (CIs) will be computed.

SECONDARY OUTCOMES:
The clinical complete remission rate (cCR) after durvalumab treatment | 36 months
  The secondary endpoints are the clinical complete remission rate (cCR) after durvalumab treatment, before surgery. The secondary end point will be assessed by means of the proportion of patients having complete remission rate (cCR) after durvalumab treatment. Corresponding two-sided 95% confidence intervals (CIs) will be computed.
Disease-free survival (DSF) | 60 months
  The disease-free survival will be evaluated during a follow up of 5 years. . DFS will be estimated by using Kaplan-Meier approach

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Degli Infermi Uo Oncologia, Faenza, Italy

REFERENCES:
- [Derived] Grassi E, Zingaretti C, Petracci E, Corbelli J, Papiani G, Banchelli I, Valli I, Frassineti GL, Passardi A, Di Bartolomeo M, Pietrantonio F, Gelsomino F, Carandina I, Banzi M, Martella L, Bonetti AV, Boccaccino A, Molinari C, Marisi G, Ugolini G, Nanni O, Tamberi S. Phase II study of capecitabine-based concomitant chemoradiation followed by durvalumab as a neoadjuvant strategy in locally advanced rectal cancer: the PANDORA trial. ESMO Open. 2023 Oct;8(5):101824. doi: 10.1016/j.esmoop.2023.101824. Epub 2023 Sep 27. PMID 37774508